CLINICAL TRIAL: NCT04111536
Title: Developing Oral LT3 Therapy For Heart Failure With Preserved Ejection Fraction
Brief Title: Developing Oral LT3 Therapy for Heart Failure - HFpEF
Acronym: DOT3HF-HFpEF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anne Cappola, MD, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 833681p; 1R61HL146390-01 (NIH)
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Low Triiodothyronine Syndrome
Keywords: Heart Failure, HFpEF, Low T3 Syndrome
MeSH Terms: conditions — Euthyroid Sick Syndromes; Heart Failure | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant, Investigators and Care Providers are blinded to LT3 vs. Placebo and T3 results. There will be 1 unblinded physician in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liothyronine (LT3), then placebo (Active Comparator): Liothyronine (L-triiodothyronine or LT3) in the 5 mcg tablet dose formulation. Minimum LT3 dose will be 2.5 mcg three times daily and the maximum LT3 dose will be 12.5 mcg three times daily.
  Interventions: Drug: liothyronine; Other: Placebo
- Placebo, then Liothyronine (Placebo Comparator): A placebo tablet matching in appearance to LT3 tablets, dosed equivalently. Minimum placebo tablet dose will be 1/2 tablet (2.5 mcg equivalent) three times daily and the maximum placebo dose will be 2 1/2 tablets (12.5 mcg equivalent) three times daily.
  Interventions: Drug: liothyronine; Other: Placebo

INTERVENTIONS:
Drug: liothyronine — Each treatment period of liothyronine was approximately 8 weeks in duration, with weekly titration of study drug for four weeks, followed by a maintenance dose for 4 weeks, then 2-week washout before crossing over to receive the alternate therapy - placebo.
  Other Names: LT3
Other: Placebo — Each treatment period of placebo was approximately 8 weeks in duration, with weekly titration of study drug for four weeks, followed by a maintenance dose for 4 weeks, then 2-week washout before crossing over to receive the alternate therapy - LT3.

SUMMARY:
Investigation of the safety, feasibility, and preliminary efficacy of thyroid hormone therapy with Liothyronine (LT3) in individuals with heart failure with preserved ejection fraction (HFpEF) and low triiodothyronine (T3) syndrome by conducting a randomized, double-blind, placebo-controlled cross-over study with a two-week washout period between treatments.

DETAILED DESCRIPTION:
The overall goal is to determine the safety, feasibility, and preliminary efficacy of administering oral LT3 therapy in the study population of participants with Heart Failure with preserved ejection fraction (HFpEF). The study will consist of two treatment periods - each treatment period will be approximately 8 weeks in duration, with weekly titration of study drug for 4 weeks, followed by a maintenance dose for 4 weeks, then 2-week washout before crossing over to the other arm (placebo or drug). LT3 will be titrated to T3 levels.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged ≥18 years; NYHA Class I, II or III heart failure or dyspnea on exertion without a clinically identifiable alternative cause; left ventricular ejection fraction greater than or equal to 40 percent; if taking antihypertensive medications, beta-blockers, SGLT2inhibitors, sacubitril/valsartan, or aldosterone antagonists, doses must be stable for at least 30 days. Elevated filling pressures as evidenced by at least 1 of the following:

1. Mitral E/e' ratio > 14 (either lateral or septal)
2. Mitral E/e' ratio > 8 (either lateral or septal), with low e' velocity (septal e'<7 cm/sec or lateral e'< 10 cm/sec), in addition to one of the following:

   1. Enlarged left atrium (LA volume index >34 ml/m2)
   2. Chronic loop diuretic use for control of symptoms
   3. Elevated natriuretic peptides (BNP levels >100 ng/L or NT-proBNP levels >300 ng/L)
   4. Tricuspid regurgitation velocity >2.8 m/s
3. Elevated invasively-determined filling pressures previously (resting LVEDP >16 mmHg or mean pulmonary capillary wedge pressure [PCWP] >12 mmHg; or PCWP/LVEDP ≥25 mmHg with exercise)
4. Acute heart failure decompensation with radiographic evidence of pulmonary venous congestion or alveolar edema, requiring IV diuretics within the past year
5. Probability of HFpEF>90%according to the HFpEF score,without a more likely apparent cause for symptoms as per Investigator assessment. TSH and free T4 level within the protocol specified reference range and total T3 level less than or equal to 0.94 ng/dL; if taking oral estrogen, dose must remain stable for duration of study participation.

Exclusion Criteria:

Hypertrophic or restrictive cardiomyopathy or uncorrected severe primary valvular disease; inability to perform VO2max exercise testing; severe lung disease; treatment with oral steroids within past 6 months for an exacerbation of obstructive lung disease, or the use of daytime oxygen; serum creatinine > 3.0 mg/dL; history of cirrhosis; acute coronary syndrome or coronary artery intervention or ablation therapy within past 2 months; cardiac surgery or percutaneous valve or septal defect repair within the past 6 months; heart failure hospitalization within past month; taking thyroid extract, LT4, LT3, amiodarone, or medication that affects the absorption or metabolism of thyroid hormone; gastrointestinal conditions that affect the absorption of thyroid hormone; current or planned pregnancy within the timeframe of study participation; any medical condition that, in the opinion of the investigator, will interfere with safe completion of the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-03-08 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne R Cappola, MD,ScM, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (8 Weeks)
Arm/Group | Liothyronine (LT3), Then Placebo | Placebo, Then Liothyronine
Started | 14 | 14
Completed | 14 | 12
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout (2 Weeks)
Arm/Group | Liothyronine (LT3), Then Placebo | Placebo, Then Liothyronine
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0
Period: Second Intervention (8 Weeks)
Arm/Group | Liothyronine (LT3), Then Placebo | Placebo, Then Liothyronine
Started | 14 | 12
Completed | 13 | 11
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liothyronine (LT3), Then Placebo | Placebo, Then Liothyronine | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 10 | 13 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 14 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Atrial Fibrillation or Ventricular Tachycardia >=4 Beats
Description: Number with atrial fibrillation or ventricular tachycardia >=4 beats
Time Frame: continuous during intervention (14 days)
Measure: Number; unit: Number of participants with events
Groups:
- Liothyronine (LT3): Participants who received liothyronine for the first 8 weeks or the last 8 weeks of the study.
- Placebo: Participants who received placebo for the first 8 weeks or the last 8 weeks of the study.
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 25 | 27
Number of participants with events | 10 | 12

2. Primary Outcome: T3 Level
Description: Number of participant T3 levels above upper limit of reference range
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 25 | 25
Participants | 7 | 0

3. Secondary Outcome: Peak Maximal Rate of Oxygen Consumption During Exercise (VO2 Max)
Description: Peak rate of oxygen consumption at 8 weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 20 | 20
ml/kg/min | 9.53 (3.42) | 10.07 (3.40)

4. Secondary Outcome: Measure of Quality of Life
Description: Change in Kansas City Cardiomyopathy Questionnaire, KCCQ scale of 0 to 100, higher score is better outcome, from baseline to 8 weeks
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | 0.1 (11.5) | 0.5 (11.1)

5. Secondary Outcome: Actigraphy
Description: Remotely sensed minutes/day of cumulative light, moderate or vigorous activity after 8 weeks of LT3 or placebo
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 24 | 25
minutes/day | 224 (70) | 230 (78)

6. Secondary Outcome: NT-proBNP Levels
Description: Change in B-type natriuretic peptide, Pg/mL, from baseline to 8 weeks
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Liothyronine (LT3) | Placebo
Number analyzed (Participants) | 25 | 25
pg/mL | 51.4 (187.6) | 8.5 (150.0)

ADVERSE EVENTS:
Time Frame: 17 weeks
Arm/Group | Liothyronine (LT3) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 2/28
Other Adverse Events (participants affected / at risk) | 10/28 | 15/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liothyronine (LT3) (N=28) | Placebo (N=28)
stroke (Vascular disorders) | 0 (0) | 1 (1)
heart failure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liothyronine (LT3) (N=28) | Placebo (N=28)
General (General disorders) | 10 (18) | 15 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT04111536/Prot_SAP_000.pdf